CLINICAL TRIAL: NCT06869642
Title: MultiCPR: The Influence of Chest Compressions on Mental Arithmetics
Acronym: MultiCPR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Mathias Maleczek, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: MultiCPR_1
Record Dates: First submitted 2025-02-25; First posted 2025-03-11 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Multitasking Behavior
MeSH Terms: conditions — Multitasking Behavior | interventions — Chest Wall Oscillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chest compression (Active Comparator): Calculations made with/without doing chest compressions - cross over design to decide what to do first, NASA-TLX will be measured
  Interventions: Behavioral: Doing Pasat-Test; Procedure: Chest compressions
- no chest compression (Active Comparator): Calculations made with/without doing chest compressions - cross over design to decide what to do first, NASA-TLX will be measured
  Interventions: Behavioral: Doing Pasat-Test

INTERVENTIONS:
Behavioral: Doing Pasat-Test — PASAT-Test either with or without doing chest compressions
Procedure: Chest compressions — Performing chest compressions as desribed in the ERC Guidelines
  Arms: Chest compression

SUMMARY:
The purpose of this clinical study is to investigate how performing chest compressions affects the ability to perform mental tasks. In particular, the effect on the participant's ability to perform mental arithmetic will be investigated. The aim is to draw conclusions about the effects of chest compressions on other mental tasks.

2 How does the clinical trial work? This clinical trial will be conducted in several locations and will involve a total of approximately 76 people in two sub-studies (38 people each). The study will be conducted by the Department of Anesthesiology of the Medical University of Vienna.

Participation in this clinical study is expected to last 30 minutes.

The following measures will be carried out exclusively for study reasons:

Depending on the sub-study you are participating in, different tasks will be performed:

Adult sub-study:

During this study, participants will be asked to perform mental arithmetic: Participants will be read a number every 2 seconds and have to add the last two in each case. The numbers are predetermined and randomly generated. At the end, we will evaluate how many results were correct.

ELIGIBILITY:
Inclusion:

* Healthy medical professionals trained in CPR (paramedics, prehospital emergency physicians, anesthesiologists, internal medicine doctors, nurses, midwifery students)
* CPR Training in the last four years
* Fit and rested.

Exclusion:

- Pregnant probands

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
PASAT Test | during the test, 2 minutes each
  Score of PAST Test

SECONDARY OUTCOMES:
Depth of chest compressions | during the pasat test, approx. 3 minutes in total
  Depth, mm
Frequency of chest compressions | during the pasat test, approx. 3 minutes in total
Leaning of chest compressions | during the pasat test, approx. 3 minutes in total
  Depth, milimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Simulation Center, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No